CLINICAL TRIAL: NCT00020852
Title: Evaluation of Freezing Tumors in the Treatment of Breast Cancer Safety Study - 1-Probe CRYOcare Surgical System for Breast Tumor Ablation
Brief Title: Cryosurgery in Treating Women With Breast Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: UCLA-9908076; CDR0000068724 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1964
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2004-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery

INTERVENTIONS:
Procedure: conventional surgery
Procedure: cryosurgery

SUMMARY:
RATIONALE: Cryosurgery kills cancer cells by freezing them. Cryosurgery followed by lumpectomy or mastectomy may be an effective treatment for breast lesions.

PURPOSE: Phase I trial to study the effectiveness of cryosurgery in treating women who have breast lesions.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of temperature-monitored, ultrasound-guided cryosurgery in women with highly suspicious breast lesions.
* Determine the safety of this procedure in these patients.

OUTLINE: This is a multicenter study.

Patients undergo cryoablation of up to two breast lesions. Within 3-21 days, patients undergo lumpectomy or mastectomy.

Patients are followed at 1, 4, 8, and 12 weeks after lumpectomy or mastectomy.

PROJECTED ACCRUAL: A maximum of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Highly suspicious breast lesion on prior mammogram and/or ultrasound with confirmation of malignancy on ultrasound-guided core biopsy

  * Tumor no greater than 2.0 cm in diameter
* Eligible for lumpectomy or mastectomy
* No superficial breast lesions
* No prior open surgical biopsy
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Any age

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics
* No other surgery that would preclude study participation

Other:

* No other medical treatment that would preclude study participation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-05; Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena R. Chang, MD, PhD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States